CLINICAL TRIAL: NCT02838264
Title: Phase 1, Open-label, Fixed Sequence, 2-period Study To Investigate The Effect Of Multiple Doses Of Itraconazole On The Pharmacokinetics Of Single Dose Pf-06463922 In Healthy Volunteers In The Fasted Condition
Brief Title: A Study To Evaluate The Effect Of Itraconazole On Pharmacokinetics Of PF-06463922 In Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Masking: None | Purpose: Basic Science
Other Study IDs: B7461012; 2016-002386-57 (EudraCT Number); ITRACONAZOLE DDI STUDY (Other: Alias Study Number)
Record Dates: First submitted 2016-07-17; First posted 2016-07-20 (Estimated); Last update posted 2017-05-15 (Actual); Status verified 2017-05

CONDITIONS: Healthy
MeSH Terms: interventions — lorlatinib; Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Cohort 1 (Experimental): All subjects in this cohort will receive the same dose of PF-06463922 in both periods. Subjects will receive PF-06463922 Alone in Period 1 followed by PF-06463922 with Itraconazole in Period 2.
  Interventions: Drug: PF-06463922; Drug: Itraconazole
- Cohort 2 (Experimental): All subjects in this cohort will receive the same dose of PF-06463922 in both periods. Subjects will receive PF-06463922 Alone in Period 1 followed by PF-06463922 with Itraconazole in Period 2.
  Interventions: Drug: PF-06463922; Drug: Itraconazole
- Cohort 3 (Experimental): All subjects in this cohort will receive the same dose of PF-06463922 in both periods. Subjects will receive PF-06463922 Alone in Period 1 followed by PF-06463922 with Itraconazole in Period 2.
  Interventions: Drug: PF-06463922; Drug: Itraconazole
- Cohort 4 (Experimental): All subjects in this cohort will receive the same dose of PF-06463922 in both periods. Subjects will receive the highest safe dose (mg) of PF-06463922 as a single-dose Alone in Period 1 followed by PF-06463922 with Itraconazole in Period 2.
  Interventions: Drug: PF-06463922; Drug: Itraconazole

INTERVENTIONS:
Drug: PF-06463922 — Single oral dose of PF-06463922 50 mg on Day 1 of Period 1 and Day 5 of Period 2
  Other Names: Lorlatinib
  Arms: Cohort 1
Drug: PF-06463922 — Single oral dose of PF-06463922 75 mg on Day 1 of Period 1 and Day 5 of Period 2
  Other Names: Lorlatinib
  Arms: Cohort 2
Drug: PF-06463922 — Single oral dose of PF-06463922 100 mg on Day 1 of Period 1 and Day 5 of Period 2
  Other Names: Lorlatinib
  Arms: Cohort 3
Drug: PF-06463922 — Highest safe single oral dose (mg) of PF-06463922 identified in the previous cohorts will be administered on Day 1 of Period 1 and Day 5 of Period 2
  Other Names: Lorlatinib
  Arms: Cohort 4
Drug: Itraconazole — 200 mg oral dose of itraconazole on Days 1 to 11 during Period 2
  Other Names: Sporanox

SUMMARY:
The purpose of this study is to estimate the effect of itraconazole on the single dose pharmacokinetics of PF-06463922 in healthy volunteers in the fasted state.

DETAILED DESCRIPTION:
This will be a Phase 1, open-label, 2-period, fixed-sequence, crossover study to investigate the effect of the strong CYP3A inhibitor itraconazole on PF-06463922 PK in approximately 16 healthy volunteers. The study will consist of potentially up to 6 treatments: single dose of PF-06463922 50, 75 or 100 mg and PF-06463922 50, 75 or 100 mg in combination with multiple dose itraconazole.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female subjects of non childbearing potential and/or male subjects, who at the time of screening, are between the ages of 18 and 55 years, inclusive.
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs).

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
* Any condition possibly affecting drug absorption.
* A positive urine drug test.
* History of HIV, Hep B or Hep C.
* History of regular alcohol consumption.
* Screening supine 12 lead ECG demonstrating PR interval >180 msec, QTc >450 msec or a QRS interval >120 msec.
* Subjects with ANY of the following abnormalities in clinical laboratory tests at screening, as assessed by the study-specific laboratory and confirmed by a single repeat, if deemed necessary: Use this criterion to describe any laboratory parameters that are not acceptable for the study. Examples included below:
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) level >1.0 × upper limit of normal (ULN);
* Total bilirubin level >1.0 × ULN; subjects with a history of Gilbert's syndrome may have direct bilirubin measured and would be eligible for this study provided the direct bilirubin level is <= ULN.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2016-08-16 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2017-05-03 (Actual)

PRIMARY OUTCOMES:
AUCinf for PF-06463922 | PF-06463922 pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and up to 168 hours post-dose.
  Area under the plasma concentration-time profile from time zero extrapolated to infinite time
Cmax for PF-06463922 | PF-06463922 pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and up to 168 hours post-dose.
  Maximum plasma concentration

SECONDARY OUTCOMES:
AUClast for PF-06463922 | PF-06463922 pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and up to 168 hours post-dose.
  Area under the plasma concentration-time profile from time zero to the time of the last quantifiable concentration (Clast)
Tmax for PF-06463922 | PF-06463922 pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and upto 168 hours post-dose.
  Time to Cmax
t1/2 for PF-06463922 | PF-06463922 pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and up to 168 hours post-dose.
  Terminal plasma elimination half-life
CL/F for PF-06463922 | PF-06463922 pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and up to 168 hours post-dose.
  Apparent clearance
Vz/F for PF-06463922 | PF-06463922 pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and up to 168 hours post-dose.
  Apparent volume of distribution
AUCinf for any potential PF-06463922 metabolite if necessary | PF-06463922 pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and up to 168 hours post-dose.
  Area under the plasma concentration-time profile from time zero extrapolated to infinite time
AUClast for any potential PF-06463922 metabolite if necessary | PF-06463922 pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and up to 168 hours post-dose.
  Area under the plasma concentration-time profile from time zero to the time of the last quantifiable concentration (Clast)
Cmax for any potential PF-06463922 metabolite if appropriate | PF-06463922 pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and up to 168 hours post-dose.
  Maximum plasma concentration
Tmax for any potential PF-06463922 metabolite if appropriate | PF-06463922 pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and up to 168 hours post-dose.
  Time to Cmax
t1/2 for any potential metabolite of PF-06463922 if appropriate | PF-06463922 pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and up to 168 hours post-dose.
  Terminal plasma elimination half-life
MRCmax for any potential PF-06463922 metabolite if appropriate | PF-06463922 pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and up to 168 hours post-dose.
  metabolite to parent ratio for Cmax
MRAUClast for any potential PF-06463922 metabolite if appropriate | PF-06463922 pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and up to 168 hours post-dose.
  metabolite to parent ratio for AUClast
MRAUCinf for any potential PF-06463922 metabolite if appropriate | PF-06463922 pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and up to 168 hours post-dose.
  metabolite to parent ratio for AUCinf
PR interval after PF-06463922 alone and after increased exposure of PF 06463922 (due to concomitant itraconzole administration). | Within 24 hours after single dose administration of PF-06463922 alone and in combination with itraconazole.
  Change in PR interval from baseline after administration of PF-06463922 single dose as assessed by ECG.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit, Brussels, Belgium

REFERENCES:
- [Derived] Patel M, Chen J, McGrory S, O'Gorman M, Nepal S, Ginman K, Pithavala YK. The effect of itraconazole on the pharmacokinetics of lorlatinib: results of a phase I, open-label, crossover study in healthy participants. Invest New Drugs. 2020 Feb;38(1):131-139. doi: 10.1007/s10637-019-00872-7. Epub 2019 Nov 14. PMID 31728714
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B7461012&StudyName=Phase+1%2C+Open-label%2C+Fixed+Sequence%2C+2-period+Study+To+Investigate+The+Effect+Of+Multiple+Doses+Of+Itraconazole+On+The+Pharmacokinetics+Of+Single+Dose+Pf-06463922+In+Healthy+Volunteers+In+The+Fasted+Condition